CLINICAL TRIAL: NCT07356115
Title: Evaluation of the Association Between PainDETECT Scores, Pain Localization, and Diagnosis in a Musculoskeletal and Sports Medicine Outpatient Population
Brief Title: Association of High PainDETECT Scores With Pain Region and Diagnosis in Patients Attending a Musculoskeletal and Sports Medicine Clinic
Acronym: PD-MSK
Status: Not yet recruiting | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Deniz Demirci, professor, Uskudar University
Other Study IDs: MSK-SPORT-PAINDETECT-01; MSK-SPORT-PAINDETECT-01 (Other: Department of Musculoskeletal and Sports Medicine, [Uskudar University ])
Record Dates: First submitted 2026-01-11; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Musculoskeletal Pain; Neuropathic Pain
Keywords: PainDETECT; Retrospective Study; Patient-Reported Outcome; Pain Assessment; Chronic Pain; Neuropathic Pain
MeSH Terms: conditions — Musculoskeletal Pain; Neuralgia; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with musculoskeletal pain: Adult patients with musculoskeletal pain whose retrospective clinical data and PainDETECT scores are analyzed.
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — This is an observational retrospective study. No interventions are assigned to participants.

SUMMARY:
This observational study aims to evaluate the relationship between PainDETECT questionnaire scores, pain regions, and clinical diagnoses in patients presenting to a musculoskeletal and sports medicine clinic. Patients attending the clinic will complete the PainDETECT questionnaire, and their pain localization and clinical diagnoses will be recorded. The findings are expected to contribute to a better understanding of neuropathic pain components in musculoskeletal conditions.

DETAILED DESCRIPTION:
This is an observational, non-interventional study conducted in a musculoskeletal and sports medicine outpatient clinic. Adult patients presenting with pain will be included. The PainDETECT questionnaire will be used to assess neuropathic pain components. Pain regions and clinical diagnoses determined during routine clinical evaluation will be recorded.

No interventions, experimental treatments, or changes to standard clinical care will be applied. The study will analyze the association between PainDETECT scores, pain localization, and clinical diagnoses. Data will be collected prospectively and analyzed using appropriate statistical methods to explore potential relationships between variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients who presented to the musculoskeletal and sports medicine clinic with pain complaints
* Availability of complete medical records including PainDETECT questionnaire data

Exclusion Criteria:

* Patients younger than 18 years
* Incomplete clinical or questionnaire data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years and older who presented to a musculoskeletal and sports medicine clinic with pain complaints and had available PainDETECT questionnaire data.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
PainDETECT Score | At baseline, based on retrospective review of existing medical records.
  The PainDETECT score is a validated patient-reported outcome measure used to assess the likelihood of neuropathic pain components. The score is calculated based on responses recorded in existing medical records. No additional assessments or interventions are performed as part of this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Cavit Meclisi - Istanbul Orthopaedics Group, Musculoskeletal and Sports Medicine Clinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the retrospective nature of the study and the absence of a predefined data sharing plan.

REFERENCES:
- [Background] Freynhagen R, Baron R, Gockel U, Tolle TR. painDETECT: a new screening questionnaire to identify neuropathic components in patients with back pain. Curr Med Res Opin. 2006 Oct;22(10):1911-20. doi: 10.1185/030079906X132488. PMID 17022849